CLINICAL TRIAL: NCT01816373
Title: Efficacy Evaluation of the Non-invasive Negative Pressure Treatment for Pectus Excavatum
Brief Title: Non-invasive Negative Pressure Treatment for Pectus Excavatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Miguel L. Tedde, MD, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDC 3591/11/009; 2011/51156-5 (Other: FAPESP)
Record Dates: First submitted 2013-03-18; First posted 2013-03-22 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Pectus Excavatum
Keywords: Chest wall; Chest, funnel; pectus excavatum; congenital abnormality
MeSH Terms: conditions — Funnel Chest; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vacuum Bell (Other): Patients with pectus excavatum will be treated with the Vacuum Bell device
  Interventions: Device: Vacuum Bell

INTERVENTIONS:
Device: Vacuum Bell — Patients with pectus excavatum will be submitted to a negative pressure treatment with the Vacuum Bell device

SUMMARY:
The purpose of this study is to determine whether the non-invasive negative pressure treatment with the use of the device Vacuum Bellfor is effective for the pectus excavatum treatment

ELIGIBILITY:
Inclusion Criteria:

* absence of co-morbidities that may interfere with proper placement or function of the apparatus
* test negative for pregnancy in women of childbearing age

Exclusion Criteria:

* skeletal diseases like osteogenesis imperfecta or osteoporosis
* clotting disorders such as hemophilia or thrombopathia
* skin diseases or infections of the anterior chest wall
* angiopathies or vascular fragility
* obesity important with BMI greater than 30
* precarious commitment to the prolonged use of the device protocol

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the reduction in the deepness of the pectus excavatum | 3 months
  The patients will be submitted to clinical measurement of their anterior chest wall at three months interval until the closing of the study

SECONDARY OUTCOMES:
Evaluation of quality of life related to self-esteem | One year
  The patients and their parents will be submitted to a quality of life questionnaire in the beginning and after one year using the device

OTHER OUTCOMES:
Evaluate the safety and adherence to the treatment | three months
  The patients will be followed to assure adherence and safety of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L. Tedde, MD, PhD, Principal Investigator — Instituto do Coracao (InCor), Hospital das Clinicas, FMUSP; Jose Ribas M de Campos, MD, PhD, Study Chair — Instituto do Coracao (InCor), Hospital das Clinicas, FMUSP
Locations (2):
- Brazil (2):
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Instituto do Coracao (InCor), Hospital das Clinicas, FMUSP, São Paulo

REFERENCES:
- [Background] Haecker FM, Sesia SB. Intraoperative use of the vacuum bell for elevating the sternum during the Nuss procedure. J Laparoendosc Adv Surg Tech A. 2012 Nov;22(9):934-6. doi: 10.1089/lap.2012.0030. PMID 23137116
- [Background] Schier F, Bahr M, Klobe E. The vacuum chest wall lifter: an innovative, nonsurgical addition to the management of pectus excavatum. J Pediatr Surg. 2005 Mar;40(3):496-500. doi: 10.1016/j.jpedsurg.2004.11.033. PMID 15793724
- [Result] Togoro SY, Tedde ML, Eisinger RS, Okumura EM, de Campos JRM, Pego-Fernandes PM. The Vacuum Bell device as a sternal lifter: An immediate effect even with a short time use. J Pediatr Surg. 2018 Mar;53(3):406-410. doi: 10.1016/j.jpedsurg.2017.04.016. Epub 2017 May 1. PMID 28495420